CLINICAL TRIAL: NCT01865799
Title: A Prospective, Observational, Drug Utilization Study of Subjects Taking Truvada for Pre-exposure Prophylaxis in the USA
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-276-0105
Record Dates: First submitted 2013-05-22; First posted 2013-05-31 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Pre-exposure Prophylaxis for Prevention of HIV Infection
Keywords: FTC/TDF; PrEP; Truvada; Drug utilization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FTC/TDF for PrEP: This prospective case series is composed of every subject in a database containing de-identified patient-level data from all healthcare channels in the US, of individuals that are exposed to FTC/TDF or its components for any indication.

SUMMARY:
This is a prospective, 3-year observational study to describe drug utilization in uninfected individuals (UIs) who initiate emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) (Truvada®) for a pre-exposure prophylaxis (PrEP) indication.

An electronic source of pharmacy/medical encounter information will be used to assess the demographics and other characteristics of the subjects prescribed FTC/TDF or its components in a prospective fashion. The data provider will supply all the de-identified information regarding each visit/interaction that the subject has had with the health system and all the diagnoses and medications that the UI has had prospectively and retrospectively for the length of time captured by the source selected.

200 physicians who prescribe FTC/TDF for a PrEP indication will be sampled from the same source.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient/ Uninfected Individual
* Adult (any sex/gender, including transgender) ≥18 years old
* Taking FTC/TDF prescribed for any indication or its components Prescriber
* Possesses an active health care professional license in good standing, with the authority to prescribe prescription medications, either independently (eg, physician) or under legally permissible arrangements for prescribing under physician supervision (eg, Nurse Practitioner or Physician Assistant)
* Practice site is within the USA
* Having prescribed FTC/TDF for a PrEP indication

Key Exclusion Criteria:

* There are no exclusion criteria for individuals or prescribers

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective case series is composed of every subject in the database that is exposed to FTC/TDF or its components for any indication.
  Additionally, 200 physicians who prescribe FTC/TDF for a PrEP indication will be randomly sampled from the same source.
Sampling Method: Non-Probability Sample
Enrollment: 64186 (Actual)
Dates: Start 2013-04-22 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Drug utilization of uninfected individuals who are prescribed FTC/TDF for a PrEP indication, including gaps in therapy | Month 36

SECONDARY OUTCOMES:
Demographics and clinical characteristics of uninfected individuals who are prescribed FTC/TDF for a PrEP indication | Months 6, 12, 18, 24, 30, and 36
  Demographics (including age, gender and if available, race and ethnicity) and clinical characteristics (including diagnoses, procedures, and laboratory test results) will be summarized by 1) exposure group and 2) overall using descriptive statistics (sample size, mean, standard deviation, median, interquartile range, minimum and maximum) for continuous data, and by the number of participants for categorical data; age will be calculated as age in years at exposure.
Demographics of prescribers of FTC/TDF for a PrEP indication | Months 6, 12, 18, 24, 30, and 36
  Demographics (including gender, medical degree, medical specialty, number of years in medical practice, and setting of care) of prescribers of FTC/TDF for a PrEP indication will be summarized using descriptive statistics (sample size, mean, standard deviation, median, interquartile range, minimum and maximum) for continuous data and by the number prescribers for categorical data.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Inc., Foster City, California, United States